CLINICAL TRIAL: NCT00525746
Title: Molecular Epidemiology of Treatment-Related Acute Myeloid Leukemia/Myelodysplastic Syndrome
Brief Title: Molecular Epidemiology of Therapy-related Acute Myeloid Leukemia/Myelodysplastic Syndrome (AML/MDS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0490
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Leukemia; MDS; AML; Malignancy; Molecular Epidemiology; Epidemiologic markers; Clinical markers; Constitutional genetic markers; Case-comparison study
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood sample collected for special tests that will look for biologic factors associated with treatment-related AML/MDS.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with a confirmed diagnosis of AML or MDS (cases).
  Interventions: Behavioral: Interview
- Controls: Patients treated for a primary malignancy (controls).
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview lasting about 50 minutes.

SUMMARY:
The goal of this research study is to identify biologic and lifestyle factors that may increase a person's risk of developing acute myeloid leukemia or myelodysplastic syndrome after treatment for a previous cancer (treatment-related AML/MDS).

DETAILED DESCRIPTION:
For this study, you will be asked to take part in a personal or mail interview. During the interview, you will be asked questions about your demographics (age, sex, etc.), any chemicals you may have been exposed to, your medical history, family history of cancer, your diet, and your smoking and alcohol use histories. It should take around 50 minutes to complete the interview. Treatment information from your medical records at M. D. Anderson will also be collected.

You will be asked to provide a saliva sample or have around 1 tablespoon of blood drawn for special tests. These tests will look for biologic factors associated with treatment-related AML/MDS.

Your participation in this study will be over once the interview has been completed and blood or saliva have been collected.

This is an investigational study. Up to 600 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Willing and able to provide written informed consent and authorization
3. Willing to donate a saliva sample or 10 ml of blood and to complete a self-administered or personal interview
4. A histologically confirmed diagnosis of AML or MDS (cases only)
5. A history of a previous primary malignancy that was treated with chemotherapy and/or radiation therapy (cases only)
6. Enrolled in leukemia/MDS studies under protocol ID00-173 or ID03-0250 (cases only)
7. Treated for a primary malignancy at MDACC (controls only)
8. Matched to cases (2:1) by cases' prior malignancy(site, treatment (chemo and/or radiation), year of diagnosis (+/- 3 years)), age (+/- 5 years), sex, and ethnicity. (controls only)

Exclusion Criteria:

1. Under 18 years of age
2. History of second primary malignancy (controls only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants, 18 years or older, with a confirmed diagnosis of AML or MDS (cases), or treated for a primary malignancy (controls).
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2006-03-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic, Clinical, + Constitutional Markers Associated with t-AML/MDS Development | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jian Gu, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org